CLINICAL TRIAL: NCT00431366
Title: The Characteristics of Sequence Effect in de Novo and Advanced Parkinson's Disease
Brief Title: Sequence Effect in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070088; 07-N-0088
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-12-24

CONDITIONS: Parkinson's Disease
Keywords: Fatigue; Repetitive TMS (rTMS); Parkinson's Disease; Peg Board Test; Levodopa; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease; Fatigue

SUMMARY:
This study will explore sequence effect, a fatigue or tiredness commonly seen in patients with Parkinson's disease after they have been doing the same thing for a while. The study will use a new device called a modified peg board test (see description below) to measure whether antiparkinsonian medications (levodopa/carbidopa or dopamine) and repetitive transcranial magnetic stimulation (rTMS, see description below) of the brain can improve the symptoms of sequence effect.

Patients with early-stage Parkinson's disease who have never taken antiparkinsonian medications and patients with advanced disease may be eligible for this study. Candidates must be 18 years of age or older and right-handed.

Participants have five visits to the NIH Clinical Center as follows:

* Visit 1 (baseline): Patients have a neurological examination, including brief cognitive function tests, a rating for depression, and two types of ratings for fatigue severity.
* Visits 2 through 5 (experimental sessions): Patients who have been taking antiparkinson medication for a long time are asked to not take their medication for about 12 hours (overnight withdrawal) before visits 2 through 5. They are off medication for about 14 hours total (until after the experiments are done). Patients may be admitted to the NIH Clinical Center for the overnight drug withdrawal if necessary. At the start of each session, participants are given either levodopa/carbidopa tablets or placebo (tablets identical in appearance but with no active medication). They perform the modified pegboard test before medication, after medication, and after brain stimulation with rTMS. During two of the sessions, they receive actual brain stimulation, and during the other two sessions they receive sham stimulation, which does not actually stimulate the brain.

The modified pegboard test is a computer-based machine with eight pegs. Subjects transfer each peg from a line of holes on the right side to a line of holes on the left side using their right hand and moving as quickly as possible. After they finish moving all pegs to the left line of holes, they wait for a beep and then transfer the pegs from left line to right line of holes. They do this six times, three times with their right hand and three times with their left.

rTMS involves repeated magnetic pulses delivered in trains or short bursts of impulses. A brief electrical current is passed through a wire coil held on the scalp. The current creates a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in muscles of the face, arm or leg. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The effect of TMS on the muscles is detected with small metal disk electrodes taped onto the skin of the right hand. Subjects receive four rTMS blocks per 10 minutes. Each block consists of a total of 375 pulses.

DETAILED DESCRIPTION:
Objective:

The long-term goal is to provide new insight into the effect of long-lasting sequence movements (sequence effect) by investigating de novo and advanced Parkinson's disease (PD) patients with an objective measurement. Our central hypothesis is that sequence effect is caused by depressed excitability of the motor cortex, and is partially associated with dopaminergic deficiency. Specifically, the aims of this study are to show that the sequence effect is more severe in advanced PD than in de novo PD and to evaluate the extent of improvement by levodopa and repetitive transcranial magnetic stimulation (rTMS) and to show the correlation of fatigue.

Study Population:

Twelve de novo PD patients and 12 age- and sex-matched advanced PD patients.

Design:

We will compare objectively measured sequence effect with a modified Purdue pegboard, a computer-based device, in de novo and advanced PD patients. The modified Purdue Pegboard will detect start and stop times for individual peg insertion and for the task in its entirety. The sequence effect in this protocol is detected by the progressive changes of time intervals per peg insertion during the testing session. A time interval is defined as the period between the start and stop times for individual peg insertion. We will conduct a placebo-controlled, four-way crossover study to determine the beneficial effect of levodopa and rTMS on the sequence effect in de novo and advanced PD. The four interventions are: levodopa and rTMS; levodopa and sham; placebo and rTMS; and placebo and sham. A replicated 4 periods and four intervention-Latin Square design will be used for the crossover design.

Outcome Measures:

The primary outcome will be the difference between two time intervals, individual 1st and 8th peg insertion time, in 1st run (8-consecutive peg insertions) with right hand, which will be compared between de novo PD and advanced PD. The secondary outcomes are: (a) the difference in progressive changes of six time values for six runs; (b) the beneficial effect of levodopa and rTMS on sequence effect; and (c) correlation between the time intervals of first and eighth peg insertion and the scores of two subjective fatigue scales, i.e., Fatigue Severity Scale (FSS) and Multidimensional Fatigue Inventory (MFI).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 years and older.
* Right hand dominant (Edinburgh Handedness Quotient greater than 60).
* Able to provide consent for the protocol.
* Hoehn & Yahr stages: I - III (de novo PD patients); II - IV (advanced PD patients).
* Never treated with antiparkinsonian medications (de novo PD patients).
* Able to go off of antiparkinsonian medications for a minimum 14 hours (advanced PD patients), i.e. overnight withdrawal until after the experiments are completed here at NIH.

EXCLUSION CRITERIA:

* Patients with any other medical, surgical, neurological or psychiatric conditions except PD.
* Patients with known symptomatic wearing off.
* Pregnant women.
* Concurrent use of tricyclic antidepressants, neuroleptic agents, or any other licit or illicit drugs other than antiparkinsonian agents that could lower the seizure threshold.
* Persons with surgically or traumatically implanted foreign bodies such as a pacemaker, an implanted medication pump, a metal plate in the skull, or metal inside the skull or eyes (other than dental appliances or fillings), intracardiac lines that may pose a physical hazard during magnetic stimulation will also be excluded.
* Patients with history of seizure disorder or epilepsy.
* Subjects without the capacity to give informed consent.
* If participation in the study would, in the opinion of the investigators, cause undue risk or stress for reasons such as excessive fatigue, general frailty, or excessive apprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2007-02-01; Study Completion 2008-12-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Patenaude H, Gelinas C, Vandal S, Fillion L. [Elaboration of a conceptual frame to explain fatigue secondary to a health difficulty and implications for nursing practice]. Rech Soins Infirm. 2002 Sep;(70):66-81. French. PMID 12385192
- [Background] Abe K, Takanashi M, Yanagihara T, Sakoda S. Pergolide mesilate may improve fatigue in patients with Parkinson's disease. Behav Neurol. 2001-2002;13(3-4):117-21. doi: 10.1155/2002/473140. PMID 12446951
- [Background] Agostino R, Berardelli A, Curra A, Accornero N, Manfredi M. Clinical impairment of sequential finger movements in Parkinson's disease. Mov Disord. 1998 May;13(3):418-21. doi: 10.1002/mds.870130308. PMID 9613731